CLINICAL TRIAL: NCT06121882
Title: A Randomized, Multi-center, Double Blind, Parallel Study to Examine the Effect of Lipogems Processed Microfragmented Adipose Tissue in Comparison to Saline for the Treatment of Knee Osteoarthritis
Brief Title: Microfragmented Adipose Tissue Compared to Saline Injection for the Treatment of Knee Osteoarthritis
Acronym: ARISE2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lipogems International spa (Industry)
Collaborators: Alira Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LIPO-002
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis; Osteo Arthritis Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor) Sponsor, Investigator, Participant are blinded. Unblinded operator will perform procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Micro Fragmented Adipose Tissue (MFat) (Experimental): Injection of Microfragmented Adipose Tissue derived using Lipogems® Kit
  The cases assigned to this group will be injected intra-articularly with Lipogems®. The patients will undergo lipoaspiration of their own adipose tissue for MFat then this MFat will be injected intra-articularly in the knee. It will be administered once at the baseline visit of the study.
  Interventions: Device: Microfragmented Adipose Tissue derived using the Lipogems® System
- Saline Injection (Active Comparator): The cases assigned to this group will be injected intra-articularly in the knee with saline. It will be administered once at the baseline visit of the study.
  Interventions: Drug: Saline Injection

INTERVENTIONS:
Device: Microfragmented Adipose Tissue derived using the Lipogems® System — Intra-articular knee injection of Microfragmented Adipose Tissue (MFat) derived using the Lipogems® System.
  Other Names: MFat
  Arms: Micro Fragmented Adipose Tissue (MFat)
Drug: Saline Injection — Intra-articular knee injection of saline
  Arms: Saline Injection

SUMMARY:
The goal of this clinical trial is to examine the effect of a single autologous, intra-articular injection of MFat versus saline injection for the treatment of pain and function associated with K/L grade 2/3 knee Osteoarthritis.

Participants will receive an injection of MFat or saline.

DETAILED DESCRIPTION:
This study will investigate The Lipogems System in a clinical study to examine the effect of adipose tissue processed using The Lipogems System in comparison to saline for the treatment of knee osteoarthritis. This study will be randomized and double-blinded. The subjects will be randomized at a 2:1 ratio (investigational to control) and will enroll 173 patients at up to 20 sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, participants must meet all of the following criteria:

  1. Age ≥ 18 years old at the date of screening
  2. Have both clinical and radiographic findings consistent with osteoarthritis of the knee:

     1. Participant has clinical findings including (but not limited to) tenderness to palpation, swelling/effusion, stiffness, chronic limited range of motion.
     2. Participant has a diagnosis of knee OA defined as Grade 2 to 3 by (K/L) weight bearing X-ray and physician review within the past 3 months.
  3. The index knee must present with symptomatic knee pain using WOMAC-A Visual Analog Scale (VAS) of 40mm or greater despite conservative therapies for 3 months prior to enrollment:

     CONFIDENTIAL Page 12 of 52 Version 2.0, 10JUL2023

     a. Failure of conservative therapies include the following: Participants must have failed a minimum of at least 3 months, including (1) physical therapy, and (2) oral OTC pain medications such as an NSAID (Aleve® or Advil®) or Acetaminophen (Tylenol®), or a prescription NSAID, for a period of 90 days at the Maximum Tolerable Dose according to the respective manufacturer's instructions on dose and duration, or their physician's over-riding guidance. Patients who are unable to tolerate this dosing regimen for 90 days, or those in whom NSAIDS or Acetaminophen are contraindicated, shall be deemed to have satisfied this inclusion criteria.
  4. Willing to give written Informed Consent to voluntarily participate in the study and sign the Health Insurance Portability and Accountability Act (HIPAA) Authorization prior to study participation
  5. Ability to return for multiple follow-up visits
  6. Ability read and understand English language
  7. Females of child-bearing potential must have a negative urine pregnancy test performed within 7 days of study enrollment or be postmenopausal (for at least 2 years) or surgically sterilized (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria:

* Participants who meet any of the following criteria will be excluded from participating in this study. Study eligibility of participants reporting isolated use of prohibited medications during the restricted periods defined by this protocol, will be evaluated on a case-by-case basis by the medical monitor.

  1. Diagnosis of knee OA defined as K/L grade 1 or 4.
  2. BMI greater than 35 kg/m2.
  3. Diagnosis of rheumatoid arthritis, psoriatic arthritis, or any other disorder which attributes to the primary source of their knee pain, including but not limited to: osteonecrosis, radiculopathy, bursitis, tendinitis, tumor, cancer.
  4. Presence of any clinically observed active infection including in the index knee joint, infection at the site of adipose tissue harvest, and/or any active systemic or local infection.
  5. Undergone injection in target knee within 6 months prior to screening visit, including but not limited to corticosteroids, hyaluronic acid (HA), bone marrow concentrate (BMAC), platelet rich plasma (PRP), human cellular exosomes, amniotic fluid, or any human birth tissue.
  6. Undergone surgical procedures of either knee within 6 months prior to the screening visit.
  7. Bilateral knee pathology can only be treated in one knee for the study. The contralateral knee must have a WOMAC-A Visual Analog Scale (VAS) pain score of no more than 20mm at the time of screening (48-hr recall).
  8. Index knee greater than 10 degrees varus/valgus deformities (anatomic tibiofemoral angle).
  9. Knee pain associated with osteochondritis dissecans, ligament damage or displaced meniscus tear.
  10. Current or historical autoimmune disease that requires immunosuppressive medication.
  11. Any disorder affecting musculoskeletal pain and/or function, including symptomatic OA of the back, hips, or ankle that would interfere with the evaluation of the treated knee.
  12. Planned or expected surgery within the next 12 months.
  13. Allergy to lidocaine, epinephrine, or valium.
  14. Diagnosis of HIV or viral hepatitis.
  15. Use of oral systemic corticosteroids within the last 90 days and for the duration of the study.
  16. History of any chemotherapy or radiation therapy of the targeted/treatment leg or adipose harvest site.
  17. Active worker's compensation case.
  18. Diagnosis of coagulation disorders (e.g., Von Willebrand's disease) and/or currently on anti-coagulant therapy.
  19. Occurrence of knee trauma to the index knee within six months prior to screening.
  20. Unwilling to stop usage of over-the-counter pain medication (e.g., Acetaminophen or NSAID), "Rescue Analgesics", for 7 days prior to any follow-up visit, with the exception of one "baby aspirin" per day for cardiovascular therapy or prophylaxis.
  21. Unwilling to stop taking prescription pain or prescription anti-inflammatory medication for the duration of the study, with the exception of Tramadol during the immediate post-procedure period noted below.
  22. Unwilling to abstain from NSAIDS for 7 days pre-injection and 2 weeks post-injection. Tramadol is allowed during the 72 hours immediately post-injection, with diary documentation of usage.
  23. Currently taking prescription pain medication for a condition other than the index knee.
  24. Currently in prison.
  25. Untreated symptomatic injury of the index knee (e.g., acute traumatic injury, anterior cruciate ligament injury, clinically symptomatic meniscus injury characterized by mechanical issue such as locking or catching).
  26. Impossibility to harvest enough adipose tissue.
  27. Any medical issue that the clinician feels would be a contraindication to the study treatment including, but not limited to:

      1. Uncontrolled diabetes defined as HbA1c >7%,
      2. History of uncontrolled hypertension defined by average systolic BP >140 mmHg or diastolic BP > 90 mmHg on ≥ 3 blood pressure medications,
      3. History of cardiovascular disease,
      4. History of cerebrovascular disease,
      5. Uncontrolled asthma, defined as symptomatic (i.e., shortness of breath and/or wheezing) despite therapy,
      6. History of solid organ or hematologic transplantation,
      7. Diagnosis of non-basal cell malignancy within preceding 5 years,
      8. Change in prescription medication within 1 month prior to enrollment,
      9. Clinically significant abnormalities in vital signs at the time of screening defined by

         * Systolic BP >140 or <90 mmHg or diastolic BP >90 or <60 mmHg
         * Pulse <55 or >100 bpm
         * Respiratory Rate <9 or >20
         * Temperature >99 °F
  28. History of septic arthritis or sepsis/bacteremia in the affected knee within 6 months prior to screening, or infection requiring antibiotic treatment within the preceding 3 months.
  29. Women who are breastfeeding.
  30. Unwilling to use contraception for 3 months post procedure unless postmenopausal (for at least 2 years) or surgically sterilized (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-06-23 (Estimated); Study Completion 2025-06-23 (Estimated)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Osteoarthritis Index Pain (WOMAC-A) VA3.1 Score | 12-month visit
  The change from baseline to Month 12 for the Western Ontario and McMaster Universities Osteoarthritis Index pain (WOMAC-A) subscale score (superiority); Scale = 0-100, where 100 is extreme pain
Change in WOMAC-C (function) Subscale Score | 12-month visit
  The change from baseline to Month 12 for the Western Ontario and McMaster Universities Osteoarthritis Index function (WOMAC-C) subscale score (non-inferiority), scale 0-100, where 100 is extreme difficulty performing a function.

SECONDARY OUTCOMES:
Change in WOMAC-A Pain Sub Score | 12-month visit
  Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC-A) Pain sub score at 6, 9 and 12-month follow-up visits compared to baseline, Scale 1-100, where 100 is extreme pain.
Change in WOMAC-C Pain Sub Score | 12-month visit
  Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC-C) Function sub score at 6, 9, and 12-month follow-up visits compared to baseline; Scale 1-100, where 100 is extreme difficulty performing a function
Change in Total WOMAC scores | 12-month visit
  Change in Total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores at, 6, 9, and 12-month follow-up visits compared to baseline; Scale 1-100, where 100 is either extreme pain (WOMAC-A), extreme stiffness (WOMAC-B) or extreme difficulty performing a function (WOMAC-C).

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Arizona Bone, Joint and Sports Medicine Center LLC, Phoenix, Arizona
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Horizon Clinical Research, La Mesa, California
  - Andrews Research & Ed Foundation, Gulf Breeze, Florida
  - Hospital for Special Surgery Florida, West Palm Beach, Florida
  - Pinnacle Trials, Inc, Atlanta, Georgia
  - Fascia Institute and Treatment (FIT) Center, Metairie, Louisiana
  - Ochsner Sports Medicine Institute, New Orleans, Louisiana
  - Regenerative Orthopedics & Sports Medicine, Rockville, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - The Orthopedic Center - NextStage Clinical Research - Tulsa, Tulsa, Oklahoma
  - LeHigh Center for Clinical Research, Allentown, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Vanderbilt Orthopaedics, Nashville, Tennessee
  - All American Ortho - NextStage Clinical Research, Houston, Texas
  - Texas Center for Cell Therapy and Research, LLC, San Antonio, Texas